CLINICAL TRIAL: NCT04211142
Title: Pain and Quality of Life After Inguinal Hernia Repair. Randomized Study Comparing Laparoscopic TAPP Repair With Open Lichtenstein Repair (QoL-TAPP Study)
Brief Title: Pain and Quality of Life After Inguinal Hernia Repair: Laparoscopic Versus Open Repair.
Acronym: QoL-TAPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QoL-TAPP
Record Dates: First submitted 2019-12-22; First posted 2019-12-26 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Hernia, Inguinal
Keywords: Hernia, Inguinal; Pain; Chronic Pain; Quality of Life; Laparoscopic Surgery; Cyanoacrylates; Mesh, Surgical
MeSH Terms: conditions — Hernia, Inguinal; Pain; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic repair (Active Comparator): Laparoscopic Transabdominal Preperitoneal Inguinal Hernia Repair (TAPP repair)
  Interventions: Procedure: Laparoscopic Transabdominal Preperitoneal Inguinal Hernia Repair (TAPP repair)
- Open repair (Active Comparator): Open Inguinal Hernia Repair (Lichtenstein repair)
  Interventions: Procedure: Open Inguinal Hernia Repair (Lichtenstein repair)

INTERVENTIONS:
Procedure: Laparoscopic Transabdominal Preperitoneal Inguinal Hernia Repair (TAPP repair) — Laparoscopic inguinal hernia repair
  Arms: Laparoscopic repair
Procedure: Open Inguinal Hernia Repair (Lichtenstein repair) — Open Inguinal Hernia Repair
  Arms: Open repair

SUMMARY:
This investigation will be a double-armed, randomized prospective study designed to compare open (Lichtenstein Technique) versus laparoscopic (TAPP) repair of primary unilateral inguinal hernia. Chronic pain, restriction of activities and esthetical outcome will be evaluated preoperatively and postoperatively, at 1, 4 and 12 months, using the European Registry for Abdominal Wall Hernias Quality of Life score (EuraHS-QoL score).

DETAILED DESCRIPTION:
Inguinal hernia repair is one of the most frequently performed surgical operations. Since the introduction of mesh repair, recurrence rates have fallen dramatically and chronic pain, as a side-effect of surgery, is becoming increasingly important.

Chronic pain is defined as pain or discomfort that lasts for more than 3 months after surgery. The reported incidence of chronic pain varies between 0 and 75 per cent after open mesh repair, and between 0 and 29 per cent after laparoscopic repair. Prospective trials suggest that there is less chronic pain after laparoscopic than open repair.

Although pain is an important parameter determining the Quality of Life (QoL) after a hernia operation, other aspects, like restriction of activities and esthetical outcome, are also of importance.

This investigation will be a double-armed, randomized prospective study designed to compare open (Lichtenstein Technique) versus laparoscopic (TAPP) repair of primary unilateral inguinal hernia.

Chronic pain, restriction of activities and esthetical outcome will be evaluated preoperatively and postoperatively, at 1, 4 and 12 months, using the European Registry for Abdominal Wall Hernias Quality of Life score (EuraHS-QoL score). The EuraHS-QoL score is a validated hernia specific questionnaire with 9 questions that can be scored by the patient in an 11-point scale from 0-10. The EuraHS-QoL questions are divided in 3 domains: "Pain" (range 0-30), "Restriction of activities" (range 0-40), and "Esthetical discomfort" (range 0-20). The total score ranges from 0-90, with the lower scores being the most favourable outcome.

The EuraHS-QoL score can be downloaded in several languages from EuraHS web pages ( http://www.eurahs.eu/EuraHS-QoL-download.php). EuraHS QoL score was previously validated and the results have been already reported in Surgery (Muysoms FE., Surgery. 2016 ;160:1344-1357)

Up to 216 patients will need to be enrolled for this study (n=108/group) and each subject will be followed for up to 12 months after the surgical intervention. The sample size was calculated to explore differences in chronic postoperative pain between the groups, accepting an α risk of 0.05 and a statistical power defined as 90 per cent (β risk = 0.1) in a two-sided test.

The study will be carried out at the Hospital Plató in Barcelona (Spain). Hospital Plató is a district general hospital serving an aggregate population of over 150.000. Hospital surgery department undertakes conventional open and laparoscopic treatment for inguinal hernia on a regular basis.

The hernia repair will be performed in all patients of both arms using the same lightweight polypropylene mesh (Optilene® 60 g/m2 ; B. Braun, Melsungen, Germany): A tailored 7.5 × 15 cm mesh for repairs in the open Lichtenstein arm, and a tailored 15 x 15 cm mesh for all patients in the laparoscopic TAPP arm. To avoid biases, meshes will be fixed in all patients (both groups) by applying liquid drops of n-butyl-2-cyanoacrylate (Histoacryl®; B. Braun Surgical, Rubí, Barcelona, Spain).

ELIGIBILITY:
Inclusion Criteria:

* primary inguinal hernia
* unilateral hernia

Exclusion Criteria:

* bilateral hernia
* recurrent hernia
* incarcerated hernia
* large scrotal hernia
* known femoral hernia
* need for associated procedures
* not able to understand the questionaire
* immunosuppression (including corticosteroids, radiotherapy, chemotherapy)
* chronic renal failure (hemodialysis)
* active infection
* pregnancy
* allergy to polypropylene or cyanoacrylate
* patient's refusal and/or absence of informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Chronic pain | 1 year
  Pain scores (0-10) using the European Registry for Abdominal Wall Hernias Quality of Life Instrument (EuraHS Quality of Life questionnaire). Each question has a scale from 0-10, whereas 0 is considered the best outcome.

SECONDARY OUTCOMES:
Restrictions of activities | 1 year
  Restrictions of activities because of pain or discomfort at the site of the hernia. Scores (0-10) using the EuraHS Quality of Life questionnaire. Each question has a scale from 0-10, whereas 0 is considered the best outcome.
Cosmetic discomfort | 1 year
  Cosmetic discomfort with abdomen shape o site of the hernia . Scores (0-10) using the EuraHS Quality of Life questionnaire. Each question has a scale from 0-10, whereas 0 is considered the best outcome.
Duration of surgery | Surgery
  Time from start of incision to skin closure
Rate of postoperative complications | 30 days
  Rate of postoperative complications (i.e., re-admission, urinary retention, symptomatic seroma, surgical-site infection). The severity of complications will be reported using the Clavien-Dindo classification system.
Early recurrences | 1-year
  Clinical recurrence or those confirmed by ultrasound examination

CONTACTS AND LOCATIONS:
Overall Officials: Salvador Guillaumes, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona; Nils Jimmy Hidalgo, MD, Principal Investigator — Hospital Clinic of Barcelona; Irene Bachero, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic, Barcelona, Spain

REFERENCES:
- [Background] Hoyuela C, Juvany M, Carvajal F, Veres A, Troyano D, Trias M, Martrat A, Ardid J, Obiols J, Lopez-Cano M. Randomized clinical trial of mesh fixation with glue or sutures for Lichtenstein hernia repair. Br J Surg. 2017 May;104(6):688-694. doi: 10.1002/bjs.10488. Epub 2017 Feb 20. PMID 28218406
- [Background] Muysoms FE, Vanlander A, Ceulemans R, Kyle-Leinhase I, Michiels M, Jacobs I, Pletinckx P, Berrevoet F. A prospective, multicenter, observational study on quality of life after laparoscopic inguinal hernia repair with ProGrip laparoscopic, self-fixating mesh according to the European Registry for Abdominal Wall Hernias Quality of Life Instrument. Surgery. 2016 Nov;160(5):1344-1357. doi: 10.1016/j.surg.2016.04.026. Epub 2016 Jun 14. PMID 27316825